CLINICAL TRIAL: NCT06821789
Title: Effects of Lacticaseibacillus Rhamnosus LRa05 on Bacterial Vaginosis and Ovarian Function in Women: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effects of Lacticaseibacillus Rhamnosus LRa05 on Bacterial Vaginosis and Ovarian Function in Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2025004
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Patients With Bacterial Vaginosis
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Conventional medication (ornidazole vaginal suppositories for 7 days) + 30B CFU/strip/day LRa05 (before meals);
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Conventional medication (ornidazole vaginal suppositories for 7 days) + maltodextrin, one strip/day (before meals);
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of this study will last 8 weeks and each subject will receive 4 follow-up visits (week 0, week 4, week 8, week 20).
  Arms: Probiotic group
Dietary Supplement: Placebo — The experimental phase of this study will last 8 weeks and each subject will receive 4 follow-up visits (week 0, week 4, week 8, week 20).
  Arms: Placebo group

SUMMARY:
In this study, Lacticaseibacillus rhamnosus LRa05 was selected as test preparations to observe the clinical efficacy in the intervention trial of combined antibiotic therapy, and to evaluate its effects on the cure rate, recurrence rate and vaginal microbiota of patients with bacterial vaginitis.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old, sexual activity, premenopausal women;
2. Nugent score for diagnosing BV ≥7;
3. Signed informed consent.

Exclusion Criteria:

1. Mixed vaginitis, such as vulvovaginal candidiasis (VVC), Trichomonas vaginalis (TV) infection, Chlamydia trachomatis (CT) infection or gonococcal vaginitis;
2. history of systemic organic disease or psychiatric illness;
3. Planning pregnancy, breastfeeding, menstruation;
4. within 5 days of the onset of the disease, any antibiotics have been used;
5. long-term use of contraceptives or immunosuppressants;
6. Allergic constitution or hypersensitivity to known components of the study drug.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Cure rate of bacterial vaginosis | 8 weeks
  The Nugent score of ≤3 is considered successful in bacterial vaginosis treatment